CLINICAL TRIAL: NCT00441220
Title: Failure of Cyclophosphamide Therapy in Lupus Nephritis Patients: the Role of Bioactivation Phenotype and Genotype
Brief Title: Cyclophosphamide in Lupus Nephritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Auckland District Health Board (Other Government); Counties Manukau Health (Other); Auckland Medical Research Foundation (Other); Arthritis New Zealand (Other)
Responsible Party: Dr Nuala Helsby, University of Auckland
Other Study IDs: ADHB3557
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Genetic polymorphisms; Cyclophosphamide; Cytochrome p450 CYP2C19 (Human); Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Patients must have lupus nephritis and previously had therapy with intravenous cyclophosphamide.
- B: Patients must have lupus nephritis and are currently receiving therapy with intravenous cyclophosphamide.

SUMMARY:
Cyclophosphamide is widely used in the treatment of cancer and autoimmune diseases such as lupus nephritis. However, there is considerable variability in the response to cyclophosphamide treatment. Cyclophosphamide is a pro-drug that requires initial activation by CYP liver enzymes. Recent clinical studies have indicated a possible role of one CYP enzyme, CYP2C19 in this activation step. This enzyme has a genetic polymorphism (variants which lack functional activity) and people who have inherited these variants are poor metabolisers of certain drugs.

The aim of this study is to determine whether response to therapy in a New Zealand population of lupus nephritis patients is determined by cyclophosphamide bioactivation (the metabolic phenotype) and CYP genotype.

Currently there is no way of predicting a patient's response to cyclophosphamide. An understanding of the factors which contribute to the therapeutic failure in lupus nephritis is particularly important due to the high morbidity and mortality associated with this disease. There are other treatment options for lupus nephritis patients who fail to respond to cyclophosphamide. If successful, this study may help identify patients who are unlikely to respond to cyclophosphamide and thus should not be unnecessarily be exposed to the drug and may justify the use of newer, more costly immunosuppressive drugs such as mycophenolate mofetil and rituximab.

DETAILED DESCRIPTION:
The autoimmune disease systemic lupus erythematosus (SLE) commonly affects the kidneys (lupus nephritis) and for some patients leads to a progressive loss of kidney function. In patients with aggressive lupus nephritis, treatment with the cytotoxic agent Cyclophosphamide (CP), and modulation of the immune system has proven effective in delaying progression of renal disease however, there is variability in how patients respond to cyclophosphamide therapy with 10% - 40% of patients failing to achieve renal remission.

Cyclophosphamide is a pro-drug, which requires metabolic bioactivation by the liver to the active drug. The major enzymes involved are CYP2C19 and CYP2B61,2 however they display considerable functional activity in part due to genetic variants which lack functional activity3. A recent study has demonstrated that lack of response to cyclophosphamide is associated with CYP2C19 and CYP2B6 poor metaboliser variants4.

A retrospective review of patients with lupus nephritis at Middlemore hospital indicated that Polynesian patients respond poorly to cyclophosphamide progressing to end stage renal failure and having higher mortality rates compared with European patients.

We have hypothesised that failure of cyclophosphamide therapy may be due to a higher incidence of the CYP2C19 variant in Polynesian populations.

An extremely high incidence (70%) of the homozygous CYP2C19 variant has been reported in the Melanesian population5 and studies in Samoan, Tongan, Cook Island and Niuean pacific peoples indicates that the incidence may be more than 4-fold higher than the 3% incidence in European populations3,6. If CYP2C19 is clinically important in the bioactivation of cyclophosphamide then Polynesian populations may be at increased risk of therapeutic failure.

Other factors may also result in inter-patient differences in the activation of cyclophosphamide in the liver. Changes in metabolic phenotype can be the result of drug-drug interactions and/or disease modulation of CYP enzyme expression. Hence it is also important to also determine the functional activity (phenotype) of cyclophosphamide bioactivation as well as genotypic analysis by analysis of blood levels of cyclophosphamide and its active metabolite.

This study will determine both the genotype and phenotype of cyclophosphamide bioactivation in patients with lupus nephritis and determine whether this is an important determinant in response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lupus nephritis requiring therapy with intravenous cyclophosphamide
* Lupus nephritis is defined according to American College of Rheumatology criteria as the presence of either:

  1. histological evidence from renal biopsy;
  2. persistent proteinuria of >0.5 g/day or proteinuria >3+ on dipstick; or
  3. cellular casts of any type. Patients will have had a renal biopsy performed to determine the histological class of lupus nephritis. Therapy with cyclophosphamide is typically used in patients with Class III, IV and severe Class V lupus nephritis.
* Patients ≥ 18 years of age
* Patients must be able to provide informed consent

Exclusion Criteria:

* Those who do not meet inclusion criteria
* Those patients in the retrospective study who have died

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lupus nephritis who are receiving or have previously received intravenous cyclophosphamide.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-10; Study Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nuala Helsby, PhD, Principal Investigator — Senior Lecturer in Molecular Medicine and Pathology, University of Auckland
Locations (3):
- New Zealand (3):
  - Auckland City Hospital, Auckland, North Island
  - University Of Auckland, Auckland
  - Middlemore Hospital, Manakau